CLINICAL TRIAL: NCT02365883
Title: Transrectal Photoacoustic Imaging of the Prostate
Status: Terminated | Type: Observational
Why Stopped: PI passed away
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-21760; PROS0044 (Other: OnCore)
Record Dates: First submitted 2015-02-11; First posted 2015-02-19 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Transrectal Imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Prostate Cancer Group
  Interventions: Device: Photoacoustic Imaging System

INTERVENTIONS:
Device: Photoacoustic Imaging System — manufactured by Endra

SUMMARY:
The purpose of this study is to image human prostate tissue using a new transrectal photoacoustic imaging probe and correlate this with ultrasound and MRI imaging performed once the specimen has been surgically removed. We hope to see what we can visualize with our device as this has never been done before. Eventually, we hope to use a similar device to image the prostate in men being seen by their doctor for prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with clinically-localized prostate cancer
* Participant desires prostatectomy
* Male
* Patient receiving treatment at Palo Alto Veterans Administration (VA) Hospital
* Age 18 to 80 years old
* English-speaking

Exclusion Criteria:

* Cannot tolerate a surgical prostatectomy due to medical comorbidities
* Cannot give informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — In order to need a prostatectomy, patient must be male.
Study Population: English-speaking men at the Palo Alto Veterans Hospital between the ages of 18 and 80 years with clinically localized prostate cancer who desire prostatectomy.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2016-12-16 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Quality of images obtained | 18 months
  Pilot study to better understand the quality of both ultrasound and photo acoustic images that can be obtained using a transrectal instrument. To understand acquisition parameters that help optimize the image quality.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv S. Gambhir, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

DOCUMENTS (1):
  • Informed Consent Form (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT02365883/ICF_000.pdf